CLINICAL TRIAL: NCT06447831
Title: Assessing Functional Capacity in Directly and Remotely Monitored Home-based Settings: A Protocol for a Multinational Validation Study in Individuals With Chronic Respiratory Diseases
Acronym: 6MST
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL) - France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-4075, 22380
Record Dates: First submitted 2024-02-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: COPD Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: Chronic Obstructive Pulmonary Disease; Exercise Capacity Test; Interstitial Lung Diseases; Physiotherapy; Rehabilitation; Telerehabilitation; Validation Study; Stepper Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lab testing (study 1): Two 3-hour laboratory visits (separated by 6 to 18 days) will be conducted. During the first laboratory visit, anthropometric measurements, pulmonary function tests and CPET on a cycle ergometer will be performed. During the second laboratory visit, spirometry will be repeated to ensure stability of the participants health state (particularly relevant for individuals with COPD). Thereafter, the 6MST and 6MWT will be performed in a randomized order, separated by a rest period of at least 30 minutes.
- At home testing (study 2): Three 1-hour home visits (separated by 2 to 5 days) will be conducted. The first trial of the 6MST (familiarization trial) will be conducted at the participant's home with the therapist present. The second and third trials of the 6MST will be performed in a randomized order, with either direct (therapist present at the home) or remote (therapist present through videoconferencing software, as in a telerehabilitation setting) monitoring.

SUMMARY:
The goal of this validation study is to provide further evidence of the metrological properties of the 6-minute stepper test in individuals with chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD).

The main questions it aims to answer are:

1. Is the 6-minute stepper test valid when compared to the 6-minute walk test and a maximal cardiopulmonary cycling test?
2. Does the 6-minute stepper test give the same results when conducted through direct (i.e., therapist in person) and remote (i.e., videoconferencing) monitoring?
3. Is the 6-minute stepper test safe when conducted at the home of the individual with direct (i.e., therapist in person) or remote (i.e., videoconferencing) monitoring?

Participants will:

* Conduct the 6-minute stepper test (several trials on separate days)
* Conduct the 6-minute walk test (1 trial on 1 day)
* Conduct a maximal cardiopulmonary test on a cycle ergometer (1 trial on 1 day)
* Participate in a semi-structured interview to provide their feedback with regards to the 6-minute stepper test

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 40 years old
* Diagnosis of chronic obstructive pulmonary disease (GOLDa 2 to 4) or of interstitial lung disease (> 6 months)
* Clinically stable for ≥ 4 weeks

Exclusion Criteria:

* Interstitial lung disease associated with connective tissue disease and sarcoidosis (often accompanied with multisystemic effects)
* Unstable or severe cardiac condition
* Invalidating rheumatologic or neurologic condition
* Weight exceeding maximal limits of exercise equipment (e.g., 130 kg for the stepper)
* Any other physical condition limiting or contraindicating exercise testing
* Simultaneous participation in another study requiring changes in medication
* Recent pulmonary rehabilitation (≤1 year, potential learning bias for the 6-minute walk test and the 6-minute stepper test)
* For arm 1 only: Use of oxygen therapy (unable to perform gas analysis with oxygen therapy)
* For arm 2 only: Participation in arm 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic obstructive pulmonary disease or interstitial lung disease followed in outpatient hospital settings
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Concurrent validity | Study 1 - Two 3-hour laboratory visits (separated by 6 to 18 days)
  Assessed using paired sample t-tests (or Wilcoxon signed-rank tests) to verify whether peak cardiorespiratory (e.g., oxygen consumption, minute ventilation, heart rate, etc.) and symptomology (i.e., dyspnea and leg fatigue) values obtained during the 6-minute stepper test are comparable to the maximal cardiopulmonary test and the 6-minute walk test
Strength of association between peak cardiorespiratory and symptomology values | Study 1 - Two 3-hour laboratory visits (separated by 6 to 18 days)
  Pearson's correlation coefficients (r) will be calculated between the number of steps taken during the 6-minute stepper test and peak oxygen consumption and heart rate reached during all three tests
Agreement | Study 1 - Two 3-hour laboratory visits (separated by 6 to 18 days)
  Assessed with Bland-Altman plots and 95% limits of agreement (mean difference ± 1.96 standard deviation of the difference) between peak cardiorespiratory and symptomology values reached during the 6-minute stepper test and those reached during the maximal cardiopulmonary test and the 6-minute walk test
Test-restest reliability | Study 2 - Trial 2 and 3 (separated by 2 to 5 days)
  Reliability (trial 2 versus 3 = directly versus remotely monitored) will be assessed using paired sample t-tests (or Wilcoxon signed-rank tests), Bland-Altman plots (with 95% limits of agreement), and intraclass correlations

SECONDARY OUTCOMES:
Adverse events | Through study completion, an average of 2 years
  All minor and serious adverse events, for all trials, will be reported
Level of comfort during test and perception of safety (qualitative) | Study 2 - Trial 3 (semi-structured interview of 20 to 30 minutes following the completion of the last trial of the 6MST)
  Assessed with thematic content analysis of semi-structured interviews (voice-recorded and transcribed)

CONTACTS AND LOCATIONS:
Locations (3):
- Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Québec, Canada
- France (2):
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, Hauts-de-France
  - FormAction Santé, Pérenchies, Hauts-de-France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bass A, Gephine S, Martin M, Belley M, Robic M, Fabre C, Grosbois JM, Dion G, Saey D, Chambellan A, Maltais F. Assessing Functional Capacity in Directly and Remotely Monitored Home-Based Settings in Individuals With Chronic Respiratory Diseases: Protocol for a Multinational Validation Study. JMIR Res Protoc. 2024 Jun 28;13:e57404. doi: 10.2196/57404. PMID 38941132